CLINICAL TRIAL: NCT01165281
Title: A Randomized, Double-Blind, Active Controlled, Optimal Dose Titration, Multicenter Study to Evaluate the Safety and Efficacy of Oral JNS024 Extended Release (ER) in Japanese and Korean Subjects With Moderate to Severe Chronic Malignant Tumor Related Cancer Pain
Brief Title: A Safety and Efficacy Study of JNS024 Extended Release (ER) in Japanese and Korean Patients With Chronic Malignant Tumor-Related Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017188; JNS024ER-KAJ-C02 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2013-12

CONDITIONS: Pain
Keywords: Pain; R331333 (JNS024ER, CG5503), tapentadol (NUCYNTA); Opioid analgesic; Oxycodone CR (OXYCONTIN CR); Chronic malignant tumor related cancer pain
MeSH Terms: conditions — Pain | interventions — Referral and Consultation; Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 001 (Experimental): R331333 (referred to as JNS024 ER or CG5503) One 25 mg to 200 mg capsule twice daily for 4 weeks.
  Interventions: Drug: R331333 (referred to as JNS024 ER or CG5503)
- 002 (Active Comparator): Oxycodone CR One 5 mg to 40 mg capsule twice daily for 4 weeks.
  Interventions: Drug: Oxycodone CR

INTERVENTIONS:
Drug: Oxycodone CR — One 5 mg to 40 mg capsule twice daily for 4 weeks.
  Arms: 002
Drug: R331333 (referred to as JNS024 ER or CG5503) — One 25 mg to 200 mg capsule twice daily for 4 weeks.
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of R331333 (referred to as JNS024 Extended-Release (ER) or CG5503) compared with an active comparator (oxycodone Controlled Release (CR)) in Japanese and Korean patients with chronic, malignant, tumor-related cancer pain.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither the patient nor the study staff will know the identity of the study drug assigned to each patient), multicenter study to evaluate the safety and efficacy of orally (by mouth) administered R331333 (referred to as JNS024 extended release [ER] capsules or CG5503) in dosages of 25 mg to 200 mg twice daily compared with orally administered capsules of oxycodone controlled release (CR) in dosages of 5 mg to 40 mg twice daily over 4 weeks in Japanese and Korean patients with moderate to severe chronic malignant tumor-related cancer pain who require around-the-clock opioid therapy (treatment with narcotic analgesics or pain relievers) and are dissatisfied with the pain relief they are experiencing from current treatment. The active control, oxycodone CR, is being used in this study because it is an opioid analgesic approved for the treatment of moderate to severe pain. Approximately 212 Japanese patients and approximately 100 Korean patients who meet screening criteria for the study will be enrolled in the study and will enter the titration period of the study where they will receive a starting dosage of either JNS024 ER 25 mg twice daily or oxycodone CR 5 mg twice daily. The dose of study drug for each patient will be titrated (increased) to the optimal dose until sufficient analgesia (pain relief) is achieved (ie, up to a maximum dose of JNS024 ER 200 mg twice daily or Oxycodone CR 40 mg twice daily). When the dosage of study drug is increased, the safety will be confirmed at the study visit or by telephone on the day after the dose is increased. Once an optimal dose of study drug is determined, the patient will continue to receive that dose during the maintenance period in the study. Patients will participate in the study for total of approximately 6 weeks; during this time patients will receive study drug for 4 weeks (titration and maintenance periods combined). During the study, if a patient experiences breakthrough pain (pain that occurs for short periods of time between doses of study drug), treatment with rescue medication (morphine immediate release [IR] 5 mg) will be given. In addition, patients will be allowed to continue to take stable doses of non-opioid analgesics (non-narcotic pain medications for mild to moderate pain) that they were taking at the time of study entry and may reduce the dosage or discontinue their use during the study. During the study, blood samples will be collected from patients at protocol-specified time points to determine the concentration of study drug after administration. The safety of patients will be monitored during the study by evaluating adverse events and findings from clinical laboratory tests, physical examinations, vital signs measurements, and electrocardiogram (ECG) measurements reported. The primary outcome measure in the study will be the change from baseline to the last 3 days of study drug administration in the average pain intensity score using an 11 point numerical rating scale (NRS). Patients will receive R331333 (referred to as JNS024 ER or CG5503) by mouth with or without food at a starting dose of 25 mg twice daily to be increased if necessary to a maximum dose of 200 mg twice daily for a total of 4 weeks (titration and maintenance periods combined) OR double-blind oxycodone CR by mouth with or without food at a starting dose of 5 mg twice daily to be increased if necessary to a maximum dose of 40 mg twice daily for a total of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical diagnosis of any type of cancer
* Diagnosis of chronic malignant tumor-related cancer pain with an average score for pain intensity in the past 24 hours of >=4 on the 11-point numerical rating scale (NRS) on the day of randomization (Day -1)
* Have not received treatment with opioid analgesics within 28 days before screening (Note: codeine phosphate [<=60 mg/d] or dihydrocodeine phosphate [<=30 mg/d] for antitussive use are allowed)
* Dissatisfied with pain relief by the current treatment and for whom the investigator or designee judges that treatment with opioid analgesics is required

Exclusion Criteria:

* Have complicated with uncontrolled/clinically significant arrhythmia
* Have previous or concurrent presence of any disease which may develop increased intracranial pressure, disturbance of consciousness, lethargy, or respiratory problems such as traumatic encephalopathy with cerebral contusion, intracranial hematoma, disturbance of consciousness, brain tumor, cerebral infarction, transient ischemic attack, epilepsy or convulsive diseases
* Have history of alcohol and/or drug abuse
* Have any disease for which opioids are contraindicated such as serious respiratory depression of serious chronic obstructive pulmonary disease, bronchial asthma attack, cardiac failure secondary to chronic pulmonary disease, paralytic ileus, status epileptics, tetanus, strychnine poisoning, acute alcohol poisoning, hypersensitivity to opium alkaloid, hemorrhagic colitis, or bacterial diarrhea

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (52):
- Japan (43):
  - Chiba
  - Fukui
  - Fukushima
  - Fukuyama
  - Fushimi
  - Hamamatsu
  - Hirosaki
  - Hitachi
  - Itami
  - Iwakuni
  - Izumo
  - Kamogawa
  - Kanuma
  - Kobe
  - Kumagaya
  - Kumamoto
  - Kure
  - Kyoto
  - Matsumoto
  - Matsusaka
  - Miyazaki
  - Nagoya
  - Natori
  - Niigata
  - Ogōri
  - Ohta
  - Okayama
  - Osaka
  - Saga
  - Saku
  - Sapporo
  - Sendai
  - Sunto
  - Takarazuka
  - Takasaki
  - Tokyo
  - Tomakomai
  - Toyama
  - Toyonaka
  - Ube
  - Yamagata
  - Yamanashi
  - Yokohama
- South Korea (9):
  - Busan
  - Chungcheongbuk-Do
  - Daegu
  - Deajun
  - Gyeonggi-do
  - Incheon
  - Jinju
  - Seoul
  - Suwon

REFERENCES:
- [Derived] Imanaka K, Tominaga Y, Etropolski M, van Hove I, Ohsaka M, Wanibe M, Hirose K, Matsumura T. Efficacy and safety of oral tapentadol extended release in Japanese and Korean patients with moderate to severe, chronic malignant tumor-related pain. Curr Med Res Opin. 2013 Oct;29(10):1399-409. doi: 10.1185/03007995.2013.831816. Epub 2013 Aug 23. PMID 23937387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To evaluate the safety and efficacy of tapentadol ER compared with oxycodone CR in Japanese and Korean patients with moderate to severe chronic cancer pain. This study was conducted from 25 Aug 2010 to 16 Aug 2012 at 69 sites in Japan and Korea. A total of 340 patients received at least 1 dose of study drug and were included in the safety analyses.
Groups:
- Tapentadol (JNS024) Extended-release (ER) Oral Tablets: Patients received tapentadol (ER) 25 to 200 mg twice daily for 4 weeks. During the titration period, the dose was titrated to the individual's optimal dose balancing efficacy and tolerability until sufficient analgesia was attained. Patients were eligible to formally enter the maintenance period if they had a pain intensity score of <=3 and did not take rescue medication more than twice daily while they were taking a stable regimen of study drug (6 identical consecutive doses) over a 3-day period. During the maintenance period, patients continued to take their optimized dose of study drug achieved during the titration period. Dosage adjustments of study drug were allowed during the titration and maintenance periods, with the exception of the last 3 days of the maintenance period when the dose was to remain unchanged.
- Oxycodone Controlled-release (CR) Oral Tablets: Patients received oxycodone controlled-release (CR) 5 to 40 mg twice daily for 4 weeks. During the titration period, the dose was titrated to the individual's optimal dose balancing efficacy and tolerability until sufficient analgesia was attained. Patients were eligible to formally enter the maintenance period if they had a pain intensity score of <=3 and did not take rescue medication more than twice daily while they were taking a stable regimen of study drug (6 identical consecutive doses) over a 3-day period. During the maintenance period, patients continued to take their optimized dose of study drug achieved during the titration period. Dosage adjustments of study drug were allowed during the titration and maintenance periods, with the exception of the last 3 days of the maintenance period when the dose was to remain unchanged.
Period: Overall Study
Arm/Group | Tapentadol (JNS024) Extended-release (ER) Oral Tablets | Oxycodone Controlled-release (CR) Oral Tablets
Started | 168 | 172
Completed | 110 | 121
Not Completed | 58 | 51
Not completed — Adverse Event | 12 | 14
Not completed — Death | 3 | 4
Not completed — Lack of Efficacy | 4 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 8 | 1
Not completed — Protocol Violation | 6 | 5
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Noncompliance with Study Drug | 1 | 4
Not completed — Progressive Disease | 10 | 14
Not completed — Other | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol (JNS024) Extended-release (ER) Oral Tablets | Oxycodone Controlled-release (CR) Oral Tablets | Total
Number analyzed (Participants) | 168 | 172 | 340
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (11.21) | 64.9 (11.41) | 65.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 72 | 150
  Male | 90 | 100 | 190
Region of Enrollment [Number; unit: participants]
  Japan | 111 | 110 | 221
  Korea | 57 | 62 | 119
Age Customized [Number; unit: Participants]
  <65 years | 77 | 79 | 156
  >=65 years | 91 | 93 | 184

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the Last 3 Days of Study Drug Administration (Last Observation Carried Forward) in the Score for Average Pain Intensity on an 11-point Numerical Rating Scale
Description: The patients recorded their average pain intensity over the past 24 hours once daily in the evening and at the same time as much as possible (eg, 10:00 PM) throughout the study in response to the following question: "What has your average pain level been for the past 24 hours, where 0=no pain and 10=pain as bad as you can imagine." The score at 3 days before the completion of study drug administration was defined as the average pain intensity score averaged over the last 3 days before completion of study drug administration.
Time Frame: Baseline, Last 3 Days of Study Drug Administration (4 weeks)
Population: Per-protocol population included all patients who were randomized, received at least 1 dose of study drug, had post-baseline efficacy data and didn't have major protocol deviations (including use of prohibited concomitant medications, non-compliance, failure to meet selection criteria, violation of regulatory requirements, or treatment deviation).
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Tapentadol (JNS024) Extended-release (ER) Oral Tablets | Oxycodone Controlled-release (CR) Oral Tablets
Number analyzed (Participants) | 126 | 139
Scores on scale | -2.69 (2.223) | -2.57 (2.027)
Statistical Analysis 1: Comparison: Tapentadol (JNS024) Extended-release (ER) Oral Tablets vs Oxycodone Controlled-release (CR) Oral Tablets; The primary hypothesis to be tested for the study was that the JNS024 ER group was not inferior to oxycodone CR as defined by the upper limit of the 95% confidence interval of the difference between JNS024 ER and oxycodone CR on the mean change from baseline of the NRS pain intensity score during the last 3 days of study drug administration. It was to be concluded that JNS024 ER is not inferior to oxycodone CR if the upper 95% confidence limit is less than 1 point; Test type: Non-Inferiority or Equivalence — In order to demonstrate that the upper limit of the confidence interval of intergroup differences in change from baseline is not higher than the noninferiority margin of 1 with a 1-tailed significance level of 0.025 and 90% power, the sample size was calculated to be 133 patients in each group for a total of 266 patients. Assuming approximately 20% of patients would be excluded from the analyses, the target sample size was 330 patients; p = 0.786, ANCOVA; Analysis of covariance (ANCOVA) model was used with treatment and country as factors and baseline pain intensity score as a covariate; Least-Squares Mean Difference = -0.06, 95% CI 2-sided [-0.506 to 0.383], Standard Error of Mean 0.226

2. Secondary Outcome: Percentage of Patients in Patient Global Impression of Change (PGIC) Score Categories
Description: The PGIC was rated by the patient and was based on the single question "Since the start of this treatment, my cancer-related pain overall is," where 1=very much improved, 2=much improved, 3=minimally improved, 4=not changed, 5=minimally worse, 6=much worse, 7=very much worse.
Time Frame: Baseline, Endpoint of the 4-week Treatment Period
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Tapentadol (JNS024) Extended-release (ER) Oral Tablets | Oxycodone Controlled-release (CR) Oral Tablets
Number analyzed (Participants) | 126 | 139
Percentage of Participants
  Percentage "much improved" or "very much improved" | 58.7 | 50.4
  Percentage "much worse" or "very much worse" | 4.0 | 1.4

3. Secondary Outcome: Frequency of Rescue Medication Use for the Double-blind Treatment Period
Description: During the study, if a patient experienced breakthrough pain (pain that occurs for short periods of time between doses of study drug), treatment with rescue medication (morphine immediate release [IR] 5 mg) was to be given. The average number of doses of Morphine IR taken per day was assessed.
Time Frame: 4 weeks
Population: This is a subset of the per-protocol population that included patients who received at least 1 dose of rescue medication. The per-protocol population included all patients who were randomized, received at least 1 dose of study drug, had post-baseline efficacy data and didn't have major protocol deviations.
Measure: Mean (Standard Deviation); unit: Number of doses per day
Arm/Group | Tapentadol (JNS024) Extended-release (ER) Oral Tablets | Oxycodone Controlled-release (CR) Oral Tablets
Number analyzed (Participants) | 94 | 103
Number of doses per day | 1.39 (0.460) | 1.35 (0.431)

4. Secondary Outcome: Total Daily Dose of Rescue Medication Use for the Double-blind Treatment Period
Description: During the study, if a patient experienced breakthrough pain (pain that occurs for short periods of time between doses of study drug), treatment with rescue medication (morphine immediate release [IR] 5 mg) was to be given. The average total daily dose of Morphine IR taken (mg) was assessed.
Time Frame: 4 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Tapentadol (JNS024) Extended-release (ER) Oral Tablets | Oxycodone Controlled-release (CR) Oral Tablets
Number analyzed (Participants) | 94 | 103
Milligrams | 6.95 (2.302) | 6.73 (2.153)

5. Secondary Outcome: Proportion of Patients With Various Levels of Pain Improvement (Responders)
Description: The proportion of patients with at least a 30 percentage improvement based on the percent change from baseline in Numerical Rating Scale score during the last 3 days of the double-blind treatment period.
Time Frame: Baseline, Last 3 Days of Study Drug Administration (4 weeks)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Tapentadol (JNS024) Extended-release (ER) Oral Tablets | Oxycodone Controlled-release (CR) Oral Tablets
Number analyzed (Participants) | 126 | 139
Percentage of Participants
  Proportion with at least a 30 percent improvement | 63.5 | 59.0
  Proportion with at least a 50 percent improvement | 50.0 | 42.4

6. Secondary Outcome: Proportion of Patients Entering the Maintenance Period
Description: Patients were eligible to formally enter the maintenance period if they had a pain intensity score of <=3 and did not take rescue medication more than twice daily while they were taking a stable regimen of study drug (6 identical consecutive doses) over a 3-day period.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Tapentadol (JNS024) Extended-release (ER) Oral Tablets | Oxycodone Controlled-release (CR) Oral Tablets
Number analyzed (Participants) | 126 | 139
Percentage of Participants | 86 | 80

7. Secondary Outcome: Number of Patients Who Discontinued Due to Lack of Efficacy
Description: The duration from the date of first study drug intake to treatment discontinuation due to lack of efficacy.
Time Frame: 4 weeks
Population: Time to discontinuation due to lack of efficacy was not analyzed since there was only 1 patient in the per-protocol set (in the tapentadol group) who discontinued treatment due to lack of efficacy.
Measure: Number; unit: Number of participants
Arm/Group | Tapentadol (JNS024) Extended-release (ER) Oral Tablets | Oxycodone Controlled-release (CR) Oral Tablets
Number analyzed (Participants) | 126 | 139
Number of participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Tapentadol (JNS024) Extended-release (ER) Oral Tablets | Oxycodone Controlled-release (CR) Oral Tablets
Serious Adverse Events (participants affected / at risk) | 78/168 | 69/172
Other Adverse Events (participants affected / at risk) | 110/168 | 127/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (JNS024) Extended-release (ER) Oral Tablets (N=168) | Oxycodone Controlled-release (CR) Oral Tablets (N=172)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Ascites (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3
Asthenia (General disorders) | 0 | 1
Disease progression (General disorders) | 40 | 36
Drug interaction (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 6
Pneumonia bacterial (Infections and infestations) | 1 | 2
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Biopsy lung (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Paralysis (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (JNS024) Extended-release (ER) Oral Tablets (N=168) | Oxycodone Controlled-release (CR) Oral Tablets (N=172)
Anaemia (Blood and lymphatic system disorders) | 4 | 11
Constipation (Gastrointestinal disorders) | 51 | 64
Diarrhoea (Gastrointestinal disorders) | 9 | 19
Nausea (Gastrointestinal disorders) | 48 | 61
Vomiting (Gastrointestinal disorders) | 41 | 41
Disease progression (General disorders) | 14 | 15
Malaise (General disorders) | 6 | 12
Pyrexia (General disorders) | 10 | 13
Decreased appetite (Metabolism and nutrition disorders) | 21 | 24
Somnolence (Nervous system disorders) | 29 | 36
Delirium (Psychiatric disorders) | 10 | 6
Insomnia (Psychiatric disorders) | 9 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. Expedited reviews will be arranged for abstracts, poster presentations, or other materials. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.